CLINICAL TRIAL: NCT04951076
Title: A Phase 2b, Randomized, Double Blind, Two Arm Study to Investigate the Effects of BNC210 Tablet Formulation Compared to Placebo in Adults With Post-Traumatic Stress Disorder (PTSD)
Brief Title: A Phase 2b Study of BNC210 Tablet Formulation in Adults With Post-Traumatic Stress Disorder (PTSD)
Acronym: ATTUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNC210.012
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNC210 (Experimental)
  Interventions: Drug: BNC210
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNC210 — BNC210 900 mg twice daily (b.i.d.) for 12 weeks
  Arms: BNC210
Drug: Placebo — Placebo twice daily (b.i.d.) for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of BNC210 compared to placebo on Post-Traumatic Stress Disorder (PTSD) symptom severity as measured by the Clinician Administered PTSD scale for The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) Total Symptom Severity Scores.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group, multi-center study with a 12 week, 2-arm treatment period. Participants will attend a Screening visit within 3 weeks before randomization to confirm eligibility. Approximately 200 participants will be randomized using a 1:1 ratio to receive either BNC210 900 mg twice daily (b.i.d.) or matched placebo. Participants will then complete 12 weeks of treatment with their allocated study intervention. Participants will return to their study site at 2-weekly intervals to complete study assessments. Participants are then requested to attend a Follow-up visit at Week 15 (i.e., 3 weeks after their last study intervention is administered).

ELIGIBILITY:
Inclusion Criteria:

* Participants with a current diagnosis of PTSD as defined by the CAPS-5 for DSM-5, with a CAPS-5 Total Symptom Severity Score of ≥30 at Screening and Baseline and no >25% decrease in Score from Screening to Baseline
* The index trauma event must have occurred in adulthood, i.e., when the participant was ≥18 years of age
* Suitable contraception use in line with protocol requirements
* Ability to swallow tablets

Exclusion Criteria:

* A period of less than 6 months since the index trauma event
* Current and ongoing exposure to the trauma that caused the PTSD
* Complex PTSD
* Severe depression as measured by a score of ≥ 35 on the Montgomery Asberg Depression Rating Scale (MADRS)
* Borderline personality disorder, bipolar disorder and other psychotic disorders
* Use of antidepressant medications within 30 days (fluoxetine within 90 days) of Screening. The use of alprazolam, flunitrazepam and chronic daily use of other benzodiazepines within 90 day of Screening.
* Failed more than three trials of antidepressant medication(s) prescribed for the treatment of PTSD.
* Concurrent trauma-based psychotherapy such as Cognitive Behavior Therapy, Prolonged Exposure Therapy, Eye Movement Desensitization and Reprocessing Therapy. Participants may however continue to receive supportive counseling that has been in place for a minimum of three months prior to Screening.
* Any moderate or severe substance use disorder in the past 12 months
* Any clinically significant medical history or findings as determined by the Investigator that could interfere with the objectives of the study or put the participant at risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (25):
  - ATTUNE Study Clinical Trial Site, Bellflower, California
  - ATTUNE Study Clinical Trial Site, Beverly Hills, California
  - ATTUNE Study Clinical Trial Site, Colton, California
  - ATTUNE Study Clinical Trial Site, Oceanside, California
  - ATTUNE Study Clinical Trial Site, Orange, California
  - ATTUNE Study Clinical Trial Site, Temecula, California
  - ATTTUNE Study Clinical Trial Site, Jacksonville, Florida
  - ATTUNE Study Clinical Trial Site, Lauderhill, Florida
  - ATTUNE Study Clinical Trial Site, Miami Lakes, Florida
  - ATTUNE Study Clinical Trial Site, Orlando, Florida
  - ATTUNE Study Clinical Trial Site, Overland Park, Kansas
  - ATTUNE Study Clinical Trial Site, Prairie Village, Kansas
  - ATTUNE Study Clinical Trial Site, New Bedford, Massachusetts
  - ATTUNE Study Clinical Trial Site, Las Vegas, Nevada
  - ATTUNE Study Clinical Trial Site, Berlin, New Jersey
  - ATTUNE Study Clinical Trial Site, Cherry Hill, New Jersey
  - ATTUNE Study Clinical Trial Site, Cedarhurst, New York
  - ATTUNE Study Clinical Trial Site, Staten Island, New York
  - ATTUNE Study Clinical Trial Site, North Canton, Ohio
  - ATTUNE Study Clinical Trial Site, Oklahoma City, Oklahoma
  - ATTUNE Study Clinical Trial Site, West Chester, Pennsylvania
  - ATTUNE Study Clinical Trial Site, Memphis, Tennessee
  - ATTUNE Study Clinical Trial Site, Austin, Texas
  - ATTUNE Study Clinical Trial Site, Dallas, Texas
  - ATTUNE Study Clinical Trial Site, Draper, Utah
- United Kingdom (7):
  - ATTUNE Study Clinical Trial Site, Barnsley
  - ATTUNE Study Clinical Trial Site, Blackpool
  - ATTUNE Study Clinical Trial Site, Cannock
  - ATTUNE Study Clinical Trial Site, Leeds
  - ATTUNE Study Clinical Trial Site, Liverpool
  - ATTUNE Study Clinical Trial Site, Manchester
  - ATTUNE Study Clinical Trial Site, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Papapetropoulos S, Doolin E, O'Connor S, Paul D, Odontiadis M, Jaros M, Rolan P, Stein MB. BNC210, an alpha7 Nicotinic Receptor Modulator, in Post-Traumatic Stress Disorder. NEJM Evid. 2025 Jan;4(1):EVIDoa2400380. doi: 10.1056/EVIDoa2400380. Epub 2024 Dec 8. PMID 39647171

RESULTS

PARTICIPANT FLOW:
Groups:
- BNC210 900 mg: BNC210 900 mg twice daily (b.i.d.) for 12 weeks
Period: Overall Study
Arm/Group | BNC210 900 mg | Placebo
Started | 106 | 106
Received Any Trial Drug | 105 | 104
Modified Intent-To-Treat (mITT) (Includes all participants who received any trial drug and had at least one post-baseline Clinician Administered Post-Traumatic Stress Disorder (PTSD) Scale for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) assessment (week 4, unless the participant completed a CAPS-5 assessment at an early termination visit between weeks 2 and 4).) | 89 | 93
Completed | 57 | 66
Not Completed | 49 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BNC210 900 mg | Placebo | Total
Number analyzed (Participants) | 105 | 104 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.01) | 42.4 (12.23) | 42.3 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 134
  Male | 40 | 35 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 24 | 50
  White | 72 | 73 | 145
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 91 | 91 | 182
  United Kingdom | 14 | 13 | 27
CAPS-5 Score [Mean (Standard Deviation); unit: Total Symptom Severity Score] — The Clinician Administered Post-Traumatic Stress Disorder (PTSD) Scale for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) is a 30-item structured interview used to diagnose PTSD and assess PTSD symptoms over the past month. Information about the frequency and intensity of each item is combined into a severity rating, and the CAPS-5 total symptom severity score is calculated by adding the severity scores for the 20 PTSD symptoms in the DSM-5. Scores range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
  Total Symptom Severity Score | 41.9 (7.51) | 41.1 (6.49) | 41.5 (7.01)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — The Clinician Global Impression - Severity (CGI-S) is a rating scale designed to assess the overall severity of the participant's symptoms. Severity is rated on a scale from 1 (normal, not at all ill) to 7 (among the most extremely ill of participants), with a higher score indicating greater severity of symptoms.
  units on a scale | 4.7 (0.64) | 4.7 (0.61) | 4.7 (0.62)
Time Since Index Trauma Event [Mean (Standard Deviation); unit: years] — Time since index trauma event occurring that caused PTSD
  years | 9.1 (9.1) | 7.9 (8.2) | 8.5 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Clinician Administered Post-Traumatic Stress Disorder (PTSD) Scale for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) Total Symptom Severity Scores After 12 Weeks
Description: The CAPS-5 is a 30-item structured interview used to diagnose PTSD and assess PTSD symptoms over the past month. Information about the frequency and intensity of each item is combined into a severity rating, and the CAPS-5 total symptom severity score is calculated by adding the severity scores for the 20 PTSD symptoms in the DSM-5. Scores range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -20.08 (1.717) | -16.05 (1.469)

2. Secondary Outcome: Change From Baseline on Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Criterion B Symptom Cluster Scores After 12 Weeks
Description: Criterion B (Intrusive Thoughts) is a 5-item sub section of the CAPS-5 scale that assesses intrusion symptoms associated with the traumatic event(s) of PTSD, with each item rated on a scale from 0 (not present) to 4 (extreme / incapacitating). Scores range from 0 to 20, with higher scores indicating greater severity of intrusion symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -5.72 (0.547) | -4.40 (0.472)

3. Secondary Outcome: Change From Baseline on Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Criterion C Symptom Cluster Scores After 12 Weeks
Description: Criterion C (Avoidance) is a 2-item sub section of the CAPS-5 scale that assesses avoidance of stimuli associated with the traumatic event(s) of PTSD, with each item rated on a scale from 0 (not present) to 4 (extreme / incapacitating). Scores range from 0 to 8, with higher scores indicating greater severity of avoidance symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -2.28 (0.299) | -1.79 (0.254)

4. Secondary Outcome: Change From Baseline on Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Criterion D Symptom Cluster Scores After 12 Weeks
Description: Criterion D (Negative Alterations in Cognitions and Mood) is a 7-item sub section of the CAPS-5 scale that assesses negative alterations in cognitions and mood associated with the traumatic event(s) of PTSD, with each item rated on a scale from 0 (not present) to 4 (extreme / incapacitating). Scores range from 0 to 28, with higher scores indicating greater severity of negative alterations in cognitions and mood symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -7.77 (0.790) | -5.98 (0.678)

5. Secondary Outcome: Change From Baseline on Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Criterion E Symptom Cluster Scores After 12 Weeks
Description: Criterion E (Arousal and Reactivity) is a 6-item sub section of the CAPS-5 scale that assesses marked alterations in arousal and reactivity associated with the traumatic event(s) of PTSD, with each item rated on a scale from 0 (not present) to 4 (extreme / incapacitating). Scores range from 0 to 24, with higher scores indicating greater severity of arousal and reactivity symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -4.35 (0.514) | -3.98 (0.436)

6. Secondary Outcome: Change From Baseline on Montgomery Asberg Depression Rating Scale (MADRS) Scores After 12 Weeks
Description: The MADRS is a 10-item clinician-rated questionnaire to measure the presence and severity of depressive episodes. Each item is rated on a scale of 0 to 6. The score from each item is combined into a total score ranging from 0 to 60, with higher scores indicating greater severity of depressive episodes.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -9.01 (1.300) | -5.82 (1.105)

7. Secondary Outcome: Change From Baseline on Hamilton Anxiety Rating Scale (HAM-A) Scores After 12 Weeks
Description: The HAM-A is an interview questionnaire that measures severity of anxiety symptoms based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior during the interview. Each parameter is rated on a scale of 0 (not present) to 4 (very severe). The score from each parameter is combined into a total score. Scores range from 0 to 56, with higher scores indicating greater severity of anxiety symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -7.10 (1.021) | -5.14 (0.875)

8. Secondary Outcome: Change From Baseline on Clinician Global Impression - Severity (CGI-S) Scale Scores After 12 Weeks
Description: The CGI-S is a rating scale designed to assess the overall severity of the participant's symptoms. Severity is rated on a scale from 1 (normal, not at all ill) to 7 (among the most extremely ill of participants), with a higher score indicating greater severity of symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -1.47 (0.173) | -1.24 (0.152)

9. Secondary Outcome: Change From Baseline on Patient Global Impression - Severity (PGI-S) Scale Scores After 12 Weeks
Description: Change from Baseline on patient-reported global functioning
  The PGI-S is a patient self-reported counterpart of the CGI-S designed to assess the patient's impression of their perceived severity of overall symptoms.Severity is rated on the PGI-S from 1 (normal) to 6 (very severe), with a higher score indicating greater severity of symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -1.25 (0.165) | -0.88 (0.144)

10. Secondary Outcome: Change From Baseline on Insomnia Severity Index (ISI) Scores After 12 Weeks
Description: The ISI is a brief self-report instrument measuring both nocturnal and diurnal symptoms of insomnia. The ISI comprises seven items, each scored from 0 to 4. The scores from each of the 7 questions are added up to get a total score of 0 to 28, with a higher score indicating a higher level of symptom severity.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -6.16 (0.906) | -3.97 (0.767)

11. Secondary Outcome: Change From Baseline on Sheehan Disability Scale (SDS) Scores After 12 Weeks
Description: The SDS is a rating scale designed to measure impairment in three domains: work/school, social life, and family life/home responsibilities. Each item is rated on a scale of 0 (not at all) to 10 (extremely), for a total score of 0 to 30, with a higher score indicating a higher degree of impairment.
Time Frame: Baseline, 4 weeks, 8 weeks,12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 93
score on a scale | -7.76 (1.033) | -6.38 (0.898)

12. Secondary Outcome: Change From Baseline on PTSD Checklist for DSM-5 (PCL-5) Scores After 12 Weeks
Description: The PCL-5 is a 20-item self-report assessment of the 20 DSM-5 symptoms of PTSD. Each symptom is rated on a scale from 0 (not at all) to 4 (extremely). Scores range from 0 to 80, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline, 12 weeks
Population: The number of participants analyzed in the placebo group differs from the total number of participants in the placebo arm in the mITT population due to a missed assessment for 1 participant at Baseline
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BNC210 900 mg | Placebo
Number analyzed (Participants) | 89 | 92
score on a scale | -21.81 (2.768) | -18.72 (2.239)

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | BNC210 900 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/105 | 2/104
Other Adverse Events (participants affected / at risk) | 36/105 | 25/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNC210 900 mg (N=105) | Placebo (N=104)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BNC210 900 mg (N=105) | Placebo (N=104)
Headache (Nervous system disorders) | 18 | 13
Nausea (Gastrointestinal disorders) | 13 | 8
Fatigue (General disorders) | 6 | 8
Eleveted Liver Enzymes (Investigations) | 14 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04951076/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04951076/SAP_001.pdf